CLINICAL TRIAL: NCT03613064
Title: Addressing Social Vulnerabilities to Prevent Hospital Readmissions in Adults With Cardiovascular Disease
Brief Title: Addressing Social Vulnerabilities in Cardiovascular Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not feasible due to local restrictions relating to COVID-19 public health emergency
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STU 022016-033; 1K23HL133441 (NIH)
Record Dates: First submitted 2018-05-31; First posted 2018-08-02 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Congestive Heart Failure; Ischemic Heart Disease; Acute Myocardial Infarction; Coronary Artery Disease
MeSH Terms: conditions — Heart Failure; Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Congestive Heart Failure (CHF) (Experimental): The CHF arm will include adults hospitalized with CHF who have been identified as being at high risk for readmission (in the top quintile of risk) by our readmission risk prediction algorithms, and who also have social vulnerabilities present. All subjects in the CHF arm will receive the Socially Enhanced Transitional Care Intervention.
  Interventions: Other: Socially Enhanced Transitional Care Intervention
- Ischemic Heart Disease (IHD) (Experimental): The IHD arm will include adults hospitalized with IHD who have been identified as being at high risk for readmission (in the top quintile of risk) by our readmission risk prediction algorithms, and who also have social vulnerabilities present. All subjects in the IHD arm will receive the Socially Enhanced Transitional Care Intervention.
  Interventions: Other: Socially Enhanced Transitional Care Intervention

INTERVENTIONS:
Other: Socially Enhanced Transitional Care Intervention — Components: 1) Standardized social vulnerabilities assessment tool, to be developed and incorporated into admission workflows. 2) Electronic community service referrals to existing community resources (i.e. food banks, shelters, community rehab), via the Dallas IEP or other information technology platform, for material (food, housing) and psychosocial needs (mental health/drug treatment). 3) Community-based cardiovascular self-management interventions, to be developed and piloted in conjunction with #3 - e.g., customized 'heart healthy' food baskets for CHF/IHD; risk factor monitoring (i.e., weight and blood pressure measurement at food banks, shelters, churches, modeled on the barber shop hypertension intervention); and 'heart buddy' support groups for CHF and IHD at community sites.

SUMMARY:
The investigators will conduct a feasibility study of an enhanced transitional care intervention, that will: 1) automate identification and risk-stratification of patients with CHF and IHD with social vulnerabilities; 2) incorporate a new standardized social vulnerabilities screening tool into clinical care; 3) enable electronic referrals to community resources; and 4) add novel community-based interventions to the existing medically-oriented transitional care intervention that is the standard of care at the study hospital (Parkland Hospital in Dallas, Texas) and other hospitals nationwide.

DETAILED DESCRIPTION:
The investigators plan to develop, pilot and evaluate the feasibility of an existing medically oriented transitional care intervention enhanced to also address social vulnerabilities, to prevent readmissions in congestive heart failure (CHF) & ischemic heart disease (IHD). The intervention design will be based on the Andersen Behavior Model of Health Services Use, highlighting pathways for clinical linkages to community resources to facilitate individual behavior change. To summarize, although existing interventions have largely focused on individual- and health system-level factors such as optimizing medication regimens, discharge education, and post-discharge follow-up, much of the risk for readmission in patients with CHF and IHD is also driven by social vulnerabilities that are currently not addressed in medical settings. Community-based organizations are a valuable but untapped resource to ameliorate key social vulnerabilities (i.e., food/housing insecurity, behavioral health needs) that are major barriers to effective medication and visit adherence, self-management and lifestyle modification in patients with heart disease. Thus, the investigators propose an enhanced transitional care intervention that uses the Dallas Information Exchange Portal, a health information technology platform, to link patients to local community organizations at discharge. Addressing social vulnerabilities to enable better adherence, self-management, and lifestyle behaviors can in turn prevent readmissions and improve downstream health outcomes. The investigators will conduct a feasibility study of an enhanced transitional care intervention, that will: 1) automate identification and risk-stratification of patients with CHF and IHD with social vulnerabilities; 2) incorporate a new standardized social vulnerabilities screening tool into clinical care; 3) enable electronic referrals to community resources; and 4) add novel community-based interventions to the existing medically-oriented transitional care intervention that is the standard of care at Parkland and other hospitals nationwide. The investigators will assess feasibility and acceptability of our intervention using measures derived from the RE-AIM (Reach, Effectiveness, Adoption, Implementation, Maintenance) implementation science framework.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized with CHF and IHD at high-risk for readmission

Exclusion Criteria:

* none

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Reach of the intervention ('R' of the RE-AIM Implementation Science Framework) | Up to 12 months
  Proportion of individuals enrolled, of those who are eligible for the intervention
Effectiveness of the intervention ('E' of the RE-AIM Implementation Science Framework) - Referrals | Up to 12 months
  Proportion of referrals to community-based service programs that are completed, of referrals that are sent. 'Completed' will be defined as individuals arriving in-person at a community-based service program after a referral is placed.
Effectiveness of the intervention ('E' of the RE-AIM Implementation Science Framework) - Health Services Utilization | Up to 12 months
  Changes in acute health services use (composite of emergency department visits, hospitalizations) before and after the intervention using interrupted time series
Effectiveness of the intervention ('E' of the RE-AIM Implementation Science Framework) - Satisfaction | Up to 12 months
  Patient satisfaction with the intervention program using brief verbal questionnaires
Adoption of the intervention ('A' of the RE-AIM Implementation Science Framework) | Up to 12 months
  Number of community organizations active in referral and information exchange intervention
Implementation of the intervention ('I' of the RE-AIM Implementation Science Framework) | Up to 12 months
  Acceptability, feasibility, and fidelity to intervention, ascertained through semi-structured interviews of research subjects, discharge planners, case managers, community program directors with thematic analysis of interview findings. We will ascertain perspectives on all three constructs during interviews and identify common themes across constructs to understand barriers and facilitators to implementation in aggregate

SECONDARY OUTCOMES:
Readmission rate | Up to 12 months
  Rate of 30-day readmissions among research subjects. We anticipate that we will be underpowered to detect a difference with our limited planned enrollment during this pilot feasibility study

CONTACTS AND LOCATIONS:
Overall Officials: Oanh K Nguyen, MD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No